CLINICAL TRIAL: NCT06112119
Title: Role of Semi-automatic MSCT Volumetry in Assessment of Rapidly Progressive Brain Atrophy in Septic ICU Patients.
Brief Title: Role of MSCT Volumetry in Assessment of Brain Atrophy in Septic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Mohamed Abdelmoneim, Assistant Lecturer, Assiut University
Other Study IDs: sepsis and brain atrophy
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Sepsis-Associated Encephalopathy
MeSH Terms: conditions — Sepsis-Associated Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- cohort: patients >16y with sepsis associated with disturbance in conscious level, the first braun CT scan will be routinely performed on admission, the second further brain CT Scan will be obtained whenever prolonged disturbance of consciousness will be detected.
  Interventions: Device: MSCT

INTERVENTIONS:
Device: MSCT — Using Semi-automatic MSCT Volumetry in assessment of brain atrophy associated with septic ICU patients

SUMMARY:
assessment of brain atrophy associated with septic ICU patients by using MSCT Volumetry

DETAILED DESCRIPTION:
Sepsis is the leading cause of admission to ICU , the number of patients who survive and discharge from ICU has also increased due to technological advances in ICU however quality of life of these patients after ICU discharge is lower than that of healthy people of a similar age, in particular Sepsis associated encephalopathy associated with brain dysfunction.

We hypothesized that brain damage including brain volume reduction that ocurre in acute phase of Sepsis using CT scan and there finding " relationship to risk factor and outcome".

We compared head CT finding at time of admission with those obtained during the course of the treatment

ELIGIBILITY:
Inclusion Criteria:

* patients >16years old with sepsis associated with disturbance in conscious level admitted to ICU

Exclusion Criteria:

* Age< 16y Brain death Hematological disease Malignant disease Hypoxemia Error in automatic tissue classification Motion artifac

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All the patients will be included within ehs inclusion criteria after giving informed consent from patients or from the hospital board to review patients' medical records, it will include:
  * Full history taking.
  * Clinically provisinal diagnosis .
  * Blood and bacterial culture was performed at the time of admission for all patients .
  * Firstly All studies were performed by using a CT device. CT scans measuring brain volume using BCR which is the width between anterior horn of the bilateral lateral ventricle divided by that of the cerebrum at the same height at the caudate nucleus that measuring in particular frontal lobe volume .
  * Also using Evan index which is the width between anterior horn of the bilateral lateral ventricles divided by cranial lumen at the same height .
  * When increase BCR and EI ,decrease in brain volume ocurr.
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
- Correlation between sepsis and brain volume reduction . - Determine the role of the CT scan in assess brain volume in acute phase of sepsis and it,s influences in improvement activities of daily living. | follow up through 10 days after admission in ICU
  - Determine the role of the CT scan in assess brain volume in acute phase of sepsis and it,s influences in improvement activities of daily living after discharge from ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Nada mohamed abdelmoneim, Principal Investigator — Assiut University; sherif mohamed abdelaal, Study Director — Assiut University; samy abdelaziz, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nakae R, Sekine T, Tagami T, Murai Y, Kodani E, Warnock G, Sato H, Morita A, Yokota H, Yokobori S. Rapidly progressive brain atrophy in septic ICU patients: a retrospective descriptive study using semiautomatic CT volumetry. Crit Care. 2021 Nov 29;25(1):411. doi: 10.1186/s13054-021-03828-7. PMID 34844648
- See also: retrospective study using semi automatic volumetry — https://doi.org/10.1186/s13054-021-03828-7